CLINICAL TRIAL: NCT03652831
Title: Effect of Soft Tissue Mobilization With and Without Neural Mobilization in Cervical Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Noor Abid, Research Associate, Isra University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIRS-IUISB/Mphil/002
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical radiculopathy,; Soft tissue mobilization,; Neural mobilization
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned randomly into two groups: Soft tissue mobilization with neural mobilization and Soft tissue mobilization without Neural mobilization.A coin will be flipped at start of data collection for the first patient to be assigned odd number and included in Soft tissue mobilization with Neural mobilization group. Later on odd and even numbered subjects will be included in specific group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft Tissues mobilization with Neural mobilization (Active Comparator): Soft Tissue Mobilization with Neural mobilization group will be assessed by spurling test and than will involved in treatment protocol i.e Cervical Traction, Hot packs, Post Isometric Relaxation Techniques and Neural mobilization Techniques which involve Median, Radial and Ulnar Nerve Mobilization.
  Frequency for neural mobilization is 3 sets of 10 repetitions for each and duration of 15minute. Participant will be scheduled to attend 12 treatment session (3 sessions every week for 4 weeks, 50mints each session)
  Interventions: Other: Soft Tissue Mobilization with Neural Mobilization
- Soft Tissues mobilization without Neural mobilization (Active Comparator): Soft Tissue Mobilization with Neural mobilization group will be assessed by spurling test and than will involved in treatment protocol i.e Cervical Traction, Hot packs, Post Isometric Relaxation Techniques.
  Participant will be scheduled to attend 12 treatment session (3 sessions every week for 4 weeks, 35mints each session)
  Interventions: Other: Soft Tissue Mobilization without Neural Mobilization

INTERVENTIONS:
Other: Soft Tissue Mobilization with Neural Mobilization — Cervical Traction for 15mints 7%of body weight with 7 second hold time and 5 second rest time.
  * Hot Pack for 10mints
  * Post isometric relaxation technique. The post-isometric relaxation technique begins by placing the muscle in a stretched position. Then an isometric contraction is exerted against minimal resistance. Relaxation and then gentle stretch follow as the muscle releases. Frequency for PIRs 3sets of 5 repetitions and duration of 10minute.
  * Neural mobilization technique includes Median, Radial and Ulnar nerve mobilization.
  Frequency for neural mobilization is 3 sets of 10 repetitions for each and duration of 15minute. Participant will be scheduled to attend 12 treatment session (3 sessions every week for 4 weeks, 50mints each session)
  Arms: Soft Tissues mobilization with Neural mobilization
Other: Soft Tissue Mobilization without Neural Mobilization — * Cervical Traction for 15mints 7%of body weight with 7 second hold time and 5 second rest time.
  * Hot Pack for 10mints
  * Post isometric relaxation technique. The post-isometric relaxation technique begins by placing the muscle in a stretched position. Then an isometric contraction is exerted against minimal resistance. Relaxation and then gentle stretch follow as the muscle releases. Frequency for PIRs 3sets of 5 repetitions and duration of 10minutes Participant will be scheduled to attend 12 treatment session (3 sessions every week for 4 weeks, 35mints each session)
  Arms: Soft Tissues mobilization without Neural mobilization

SUMMARY:
This study will evaluate effect of soft tissue mobilization with and with out neural mobilization in cervical radiculopathy, half of the subjects will receive treatment of soft tissue mobilization along with neural mobilization whereas half of the subjects will receive only soft tissue mobilization.

DETAILED DESCRIPTION:
soft tissue mobilization and neural mobilization both treatments are used to treat cervical radiculopathy but they work differently.

Soft tissue mobilization include traction which decompresses the nerve and stretches the surrounding muscles along with help to reduce pain and tingling sensation. whereas hot pack helps to increase blood circulation and warm up muscles and isometric exercises provide strengthening and build endurance.

Neural mobilization technique is different for all 3 nerves i.e Radial, ulnar and median. neural mobilization technique target the single nerve which is being compressed and showing symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age 18 to 55years
* Patients having pain more than 3months
* Radiating pain in one of the upper limb
* Spurling's test positive

Exclusion Criteria:

* Traumatic injury of upper limb or cervical spine
* Vertebral artery test positive(dizziness, vomiting, diplopia, drop attacks etc)
* Patient asymptomatic for pain but symptomatic for tingling and paraesthesia
* Circulatory disturbance of upper extremity
* Known history of high level of spinal cord injury and malignancy
* Thoracic Outlet syndrome

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4weeks
  Pain intensity in one of the upper limb is measured by Numeric pain scale in which "0" shows No pain while "10" shows worst pain.

SECONDARY OUTCOMES:
Recurrence of pain and Neck disability | 4weeks
  Neck disability index scale used to measure ability to manage neck pain in everyday life in terms of: Pain intensity, Personal care, Lifting, Reading, Headaches, and Concentration. In which "0" shows disability and "5" shows normal.
Neck Range of Motion | 4weeks
  Range of motion of the cervical spine and upper extremity (any of the upper limb) measured by Goniometer. Values deviated from standard values are considered as abnormal. The DASH Outcome Measure is scored as: the disability/symptom section (30 items, scored 1-5) where "1" shows No difficulty and "5" shows maximal difficulty

IPD SHARING:
Plan to Share IPD: Undecided